CLINICAL TRIAL: NCT00213837
Title: Reconstruction Implant Bone (Anterior Mandibular Arch) After Removing Using Porous Titanium Prosthesis in ENT Surgery
Brief Title: Reconstruction Implant Bone After Removal Using Porous Titanium Prosthesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3096
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Otorhinolaryngologic Diseases
Keywords: porous titanium implants; thyroplasty; vocal cord paralysis; male or female more than 18 years old
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Vocal Cord Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Mandibular prosthesis made of a new highly biointegratable material — Replacement of mandibular bone after partial or total mandible resection,avoiding then bone grafting. The porous titanium prosthesis is implanted under general anaesthesia in laryngeal surgeries. Bone resection and prosthesis placement is performed during the same surgical intervention. The prosthesis is attached onto the healthy bone with surgical screws. Simultaneous grafting of vascularised tissues may be done if the prosthesis surrounding area has been strongly irradiated.

SUMMARY:
This trial will study the reconstruction of the anterior part of the mandible and the adjacent soft tissue parts by a mandibular prosthesis made in porous titanium, associated or not, to a latissimus dorsi or pectoral flap, to avoid reconstruction with free microanastomosed bone flaps that are often associated with important morbidity.

The implant is consolidated by two prolonged parallel plates of titanium, allowing their fixation to the bone, easy to fix in a short time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female more than 18 years old

Exclusion Criteria:

* Age less than 18 years old
* Pregnant women
* Local carcinoma excluding radiotherapic or surgical control
* Poor general condition
* Contraindication to general anesthesia
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
TEP scan + MRI + CT scan | 3 months after surgery
Blood analysis (interleukin) | 8, 15, 30 days and 3 months after surgery
All types of complication | 8, 15, 30 days, 3, 6 months after surgery and then every 6 months during the whole trial

CONTACTS AND LOCATIONS:
Overall Officials: Christian Debry, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Service d'Oto-Rhino-Laryngologie et de Chirurgie Cervico-Faciale, Hôpital de Hautepierre, Strasbourg, France

REFERENCES:
- [Result] Schultz P, Vautier D, Atallah I, Gentine A, Debry C. [Reconstruction of the anterior mandibule using a porous titanium implant: a case report]. Rev Laryngol Otol Rhinol (Bord). 2008;129(3):201-5. French. PMID 19694164